CLINICAL TRIAL: NCT04945408
Title: Longitudinal Description of Hemorrhoidal Pathology
Acronym: DeLPH
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DeLPH Cohort
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2022-03

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemorrhoidal disease is a common cause of gastroenterology visits. In the United States, it is considered the 3rd most common gastrointestinal diagnosis with nearly 4 million scheduled or emergency visits. In France, self-reported questionnaires estimate that one person in five has suffered at least one hemorrhoidal attack in the past year.

DETAILED DESCRIPTION:
Hemorrhoidal disease significantly alters the quality of life, can be life threatening in case of heavy bleeding and has a significant economic impact.

However, there are still many unknowns regarding the different types of hemorrhoidal disease, its symptoms, its natural history, its etiology, its triggering and promoting factors, the associated pathologies, the therapeutic indications, etc.

In addition, the therapeutic management is not consensual, especially since the therapeutic arsenal is constantly expanding over the last 20 years with the advent of minimally invasive surgical techniques.

The aim of the work is to answer some of these questions on the basis of a prospective cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Consecutive patients consulting for hemorrhoidal disease at the proctology department of the Groupe Hospitalier Paris Saint-Joseph (GHPSJ) between January 1, 2020 and April 30, 2020
* French-speaking patient

Exclusion Criteria:

* Patient objecting to participation in the study
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients consulting for hemorrhoidal disease in the proctology department of the Groupe Hospitalier Paris Saint-Joseph (GHPSJ) between January 1st 2020 and April 30th 2020
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the different treatments proposed according to the type of hemorrhoidal disease (internal, external or both) | 6 months
  Average prolapse score before and after treatment according to the type of hemorrhoidal disease (internal, external or both).
Evaluate the effectiveness of the different treatments proposed according to the type of hemorrhoidal disease (internal, external or both) | 6 months
  Average bleeding score before and after treatment according to the type of hemorrhoidal disease (internal, external or both).
Evaluate the effectiveness of the different treatments proposed according to the type of hemorrhoidal disease (internal, external or both) | 6 months
  Average quality of life score before and after treatment according to the type of hemorrhoidal disease (internal, external or both).

SECONDARY OUTCOMES:
Evaluate the proportion of patients consulting for hemorrhoidal disease in the general proctology consultation of a specialized center that also receives emergencies | 6 months
  Proportion of patients in the proctology department consulting for hemorrhoidal disease
Describe the various symptoms of hemorrhoidal disease | 6 months
  Proportions of various symptoms of hemorrhoidal disease
Search for proctological pathologies associated with hemorrhoidal disease | 6 months
  Prevalence of proctological pathologies associated with hemorrhoidal disease
Determine potential risk factors for hemorrhoidal disease | 6 months
  Correlations between potential risk factors and the development of hemorrhoidal disease

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France